CLINICAL TRIAL: NCT01944189
Title: Artemether/ Lumefantrine: A Study of the Effect of Local Food on Pharmacokinetics of Lumefantrine and Population Pharmacokinetics of Lumefantrine Among Ugandan Children
Brief Title: Artemether/ Lumefantrine: A Study of the Effect of Local Food on Pharmacokinetics and Population Pharmacokinetics
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makerere University (Other)
Collaborators: Karolinska Institutet (Other); Swedish International Development Cooperation Agency (SIDA) (Other Government)
Responsible Party: Principal Investigator, College of Health Sciences, Dr Norah Mwebaza, Makerere University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: HS 567; 2009/054 (Other: Makerere University Research Ethics Committee)
Record Dates: First submitted 2013-09-04; First posted 2013-09-17 (Estimated); Last update posted 2014-05-28 (Estimated); Status verified 2014-05

CONDITIONS: Malaria, Falciparum
Keywords: lumefantrine pharmacokinetics & bioavailability
MeSH Terms: conditions — Malaria, Falciparum | interventions — Food; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Food Supplement (Experimental): Population PK Study will enroll 70 children receiving standard AL dose at 0, 8, 24, 36, 48, 60 hour with recommended milk or maize porridge plus oil. Both foods contain sufficient fat therefore will contribute to pool evaluations as a single cohort.
  A subset, 48 children will have participated in nested comparative bio-availability study as follows Standard arm children receiving single dose with milk (12) Standard arm children receiving double dose with milk (12) Experimental arm children receiving single dose with maize porridge plus oil (12) Experimental arm children receiving double dose with maize porridge plus oil (12) The rest, 22 children will have participated exclusively in PPK, receiving appropriate single or double dose with milk similar to those in standard arm
  Interventions: Dietary Supplement: Food
- Food Supplement Arm (Experimental): Population PK Study will enroll 70 children receiving standard AL dose at 0, 8, 24, 36, 48, 60 hour with recommended milk or maize porridge plus oil. Both foods contain sufficient fat therefore will contribute to pool evaluations as a single cohort.
  A subset, 48 children will have participated in nested comparative bio-availability study as follows Standard arm children receiving single dose with milk (12) Standard arm children receiving double dose with milk (12) Experimental arm children receiving single dose with maize porridge plus oil (12) Experimental arm children receiving double dose with maize porridge plus oil (12) The rest, 22 children will have participated exclusively in PPK, receiving appropriate single or double dose with milk similar to those in standard arm
  Interventions: Dietary Supplement: Food

INTERVENTIONS:
Dietary Supplement: Food — Nested comparative bioavailability study: 48 out of 70 children randomized to 2 food arms under 2 dose groups of artemether lumefantrine (20mg /120 mg) treatment according to standard care weight based dose groups (> 5 to >15 kg receive 1 tablet and 15 to > 25 kg receive 2 tablets)
  Food arms:
  Standard arm = Milk
  Experimental arm = maize porridge plus oil
  Groups include Single dose group= 1 tablet of artemether lumefantrine (20/120 mg) and Double dose group= 2 tablet of artemether lumefantrine (20/120 mg)
  Standard arm children receiving milk and single dose(12) Standard arm children receiving milk and double dose(12) Experimental arm children receiving maize porridge plus oil and single dose(12) Experimental arm children receiving maize porridge plus oil and double dose (12)
  Other Names: Coartem Dispersible 20/120 mg; NAFDAC REG.NO.: A4-1680

SUMMARY:
Despite preventive programs, effective case management is still the cornerstone in malaria control.

This study is as a strategy towards improved recommendations in resource limited countries during artemether -lumefantrine (AL) treatment in order to maximize the public health benefits.

This is observational population pharmacokinetics study with a nested comparative bioavailability study.The study is intended to describe the variability in lumefantrine blood levels among under five year old Ugandan children with uncomplicated falciparum malaria receiving current standard artemether-lumefantrine dose regimens. Findings will form a basis for development of rational dosage recommendations. The nested comparative bioavailability study will explore effect of profiled local food intake (maize porridge plus vegetable oil versus milk) on lumefantrine uptake. As a strategy towards improved recommendations in resource limited countries during AL treatment in order to maximize the public health benefits. As a secondary objective we will correlate the variability in lumefantrine uptake to malaria treatment outcome and safety profile in this population.

Research hypotheses

1. The population pharmacokinetic profile of lumefantrine among under five year old children in Uganda with uncomplicated falciparum malaria is not affected by demographic factors.
2. There is no difference in the bioavailability of lumefantrine when artemether-lumefantrine is received with maize porridge plus vegetable oil versus milk among under five year old Ugandan children treated for uncomplicated falciparum malaria.

DETAILED DESCRIPTION:
This is an observational study with a nested comparative bioavailability study among children based at Mulago Hospital, Kampala Uganda. It is a part of profiled doctoral study project aimed at improving artemether-lumefantrine drug use among children in resource limited settings in order to maximize public health benefits. It involves initial healthy volunteer studies, quantitative analytical studies and finally this pediatric patient study.

Artemether-lumefantrine is currently the first line treatment of uncomplicated malaria in Uganda and several countries in sub Saharan Africa. Currently the recommended dose regimens for children, the most vulnerable population are still empirically weight based derivations based on mainly clinical experience from studies done among adults. Yet children are physiologically different from adults. In particular lumefantrine, a long acting agent ensuring radical cure is highly lipophilic, and has variable oral bioavailability. High variability of lumefantrine uptake and its long half life render it liable to selection pressure if sub-therapeutic concentrations prevail for long periods. Recommended milk or high fat diet to improve its bioavailability may not be available in resource limited settings. In Mwebaza et al ., 2013, our health volunteer crossover bioavailability study preceding the planned patients study, lumefantrine exposure was comparable in milk and maize porridge plus oil study groups. Whereas both fasted and maize porridge groups demonstrated similarly much lower ranges of lumefantrine exposures relative to milk. The greatly improved absorption is attributed to the little fat used to fortify maize porridge. We believe that findings in healthy adult volunteers are relevant for vulnerable African children treated with AL for P. falciparum malaria but this needs to be confirmed.

Objectives

1. To describe the population pharmacokinetics of lumefantrine among under five year old children in Uganda receiving AL for uncomplicated falciparum malaria (Main study).

   The described PPK profile will be correlated to treatment outcomes and will form a basis for dose recommendations.
2. To compare the effects of maize porridge plus vegetable oil versus milk on the bioavailability of lumefantrine among under five year old Ugandan children receiving artemether- lumefantrine for uncomplicated falciparum malaria (Nested Study).

This study will establish whether it is possible to recommend fortification of carbohydrate rich food with little fat (maize porridge plus vegetable oil) to achieve similarly optimal absorption of lumefantrine , if milk is not available in resource limited setting during artemether lumefantrine treatment for uncomplicated malaria.

Mani sub-study (1). A single centre open-label prospective non-comparative pharmacokinetic study will be carried out at the Department of Pharmacology & Therapeutics, Makerere University College of Health Sciences, at Mulago Hospital Complex, Kampala, Uganda. Study will include children (less than 5 years, n=70) diagnosed with uncomplicated falciparum malaria destined to receive standard fixed-weight-based six-dose regimen of artemether-lumefantrine for 3 days on outpatient basis . A full population pharmacokinetic design will be employed to obtain sparse venous plasma samples from participants at scheduled periods during a 28 day follow up period. Each participant will provide between 1 to 8 samples during the 28 day follow up period. Venous plasma levels of lumefantrine (L) and its metabolite desbutyl-lumefantrine (DL) will be determined using liquid chromatography and mass spectrometry tandem (LCMS/MS) at the Division of Clinical Pharmacology, Department of Laboratory Medicine, Karolinska Institute, Stockholm, Sweden. Outcome variables will be pharmacokinetic (PK) exposure parameters of L and DL. Sparse PK data will be pooled for evaluation of both individual and population PK parameter estimates of lumefantrine using NONMEM. Impact of patients' explanatory variables on PK parameters will be assessed. Secondary outcomes will include be adverse events and day 28 treatment outcome.

Nested sub-study (2), is a comparative bioavailability study to compare lumefantrine bioavailability after the first oral dose of AL among pediatric patients receiving standard care. Forty eight out of the 70 under five year old children with uncomplicated malaria will be randomized to receive AL with either milk (n=24) or local maize porridge plus oil (n=24). Venous plasma concentrations (1 ml, whole blood) will be obtained up to 8 hours (at 0, 1, 1.5, 2, 3, 4, 6, 8) after the first using an intensive pharmacokinetic sampling design. Thereafter 1 to 8 sparse venous blood samples will be obtained during a 28 day follow up period to contribute to the PPK study pool. Primary Pharmacokinetic endpoints and outcomes will be exposure parameters after first dose, up to 8 h. Peak concentrations (Cmax) and early exposure (AUC0-8h) will be used for relative bioavailability evaluations using confidence interval approach for average bioequivalence. Secondary end points will be day 28 in follow up with lumefantrine PK exposure (AUC0-28d and AUC0-∞) and day 28 treatment outcomes as secondary outcomes. Correlation of overall exposure (AUC0-28d and AUC0-∞) to clinical and parasitological response to AL treatment will be explored.

ELIGIBILITY:
Inclusion criteria:

* Diagnosis of uncomplicated falciparum malaria
* Age ≥ 6 months to ≤5 years.
* For nested comparative bioavailability study, age >1 to ≤5 years of age, to avoid intense blood draws from younger children
* Weight ≥5 kg.
* For nested comparative bioavailability study, restrict evaluation to 2 weight/dose groups >5 to < 15kg and 15 to < 25kg
* Within 10 km radius from recruitment site
* Informed consent from parent or guardian
* Willingness to adherence to study procedures

Exclusion criteria:

* Severe or complicated malaria "Danger signs"
* Mixed plasmodial infection
* Hemoglobin < 5 mg/dl
* Weight < 5kg
* Allergy to study medication or milk
* Medication which known to inhibit or induce CYP3A4/5 examples ketoconazole, erythromycin, steroids, antidepressants, anticonvulsants, antiretroviral drugs.
* Receipt of artemisinin containing compounds in the past 7 days or lumefantrine in the past 28 days

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-09 (Estimated); Study Completion 2015-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic (PK) exposure parameters of lumefantrine | 28 days
  Sparse pharmacokinetic data will be pooled for evaluation of both individual and population PK parameter estimates of lumefantrine using Non linear mixed effect model. Pharmacokinetic exposure will be depicted principally by area under the concentration-time curves following the last dose through to 28 days of follow up (AUC0-28). Other PK parameters portraying exposure will also be assessed alongside. These include half life (t1/2), peak concentrations (Cmax) and time to reach Cmax (Tmax), apparent clearance and volumes of distribution.

SECONDARY OUTCOMES:
Relative Oral Bioavailability of lumefantrine | 8 h after the first dose
  Nested Randomized Comparative Bioavailability study: Relative oral bioavailability between the two food arms will be assessed using lumefantrine pharmacokinetic exposure outcomes at 8 h after first dose. Parameters to be considered will be attained peak concentrations (Cmax ) and area under concentration-time curve up to 8h after the first dose (AUC0-8h).
  Peak concentrations (Cmax) and AUC0-8h will be used for relative bioavailability evaluations using confidence interval approach for average bioequivalence.

OTHER OUTCOMES:
Malaria treatment outcome (clinical and parasitological response) | 28 days
  Correlation of overall lumefantrine exposure (AUC0-28d and AUC0-∞) to clinical and parasitological response to artemether lumefantrine treatment will be explored.
Adverse events | 28 days
  To assess the relationship between drug exposure over the time and the safety profile in particular clinical parameters

CONTACTS AND LOCATIONS:
Overall Officials: Norah Mwebaza, MBChB M Sc, Principal Investigator — • Department of Pharmacology and Therapeutics, Makerere University College of Health Sciences (MakCHS), Uganda; Urban Hellgren, MD PhD, Study Chair — Div Infectious Diseases, Karolinska Institutet (KI) , Sweden; Lars L Gustaffson, MD PhD, Study Chair — Dep Lab Medicine, Div Clinical Pharmacology, KI; Paul Waako, PhD, Study Chair — Department of Pharmacology and Therapeutics, MakCHS, Kampala, Uganda; Celestino Obua, PhD, Study Chair — Department of Pharmacology and Therapeutics, MakCHS, Kampala, Uganda
Locations (1):
- Department of Pharmacology & Therapeutics, MakCHS, Mulago Hospital Complex, Kampala, Uganda

REFERENCES:
- [Background] Mwebaza N, Jerling M, Gustafsson LL, Obua C, Waako P, Mahindi M, Ntale M, Beck O, Hellgren U. Comparable lumefantrine oral bioavailability when co-administered with oil-fortified maize porridge or milk in healthy volunteers. Basic Clin Pharmacol Toxicol. 2013 Jul;113(1):66-72. doi: 10.1111/bcpt.12065. Epub 2013 Apr 6. PMID 23480875